CLINICAL TRIAL: NCT00680602
Title: Group Cognitive Behavioral Therapy Versus Fluoxetine for Obsessive-Compulsive Disorder: a Randomized Open Trial for Any Patient.
Brief Title: Group Cognitive Behavioral Therapy Versus Fluoxetine for Obsessive-Compulsive Disorder: a Practical Trial
Acronym: GCBTVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Cristina Belotto da Silva, Department & Institute of Psychiatry, Clinical Hospital, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 06/50829-8
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Obsessive Compulsive Disorder
Keywords: behavior therapy; group therapy; psychopharmacology
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Behavior Therapy; Psychotherapy, Group; Selective Serotonin Reuptake Inhibitors; Fluoxetine; Sertraline; Paroxetine; Citalopram; Dexetimide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Group Cognitive Behavior Therapy
  Interventions: Behavioral: Group Cognitive Behavior Therapy
- 2 (Active Comparator): Selective Serotonin Reuptake Inhibitor
  Interventions: Drug: SSRI (fluoxetine, sertraline, paroxetine, citalopram)

INTERVENTIONS:
Behavioral: Group Cognitive Behavior Therapy — Structured protocol described by Cordioli et al., 2003
  Other Names: behavior therapy; CBT; group psychotherapy
  Arms: 1
Drug: SSRI (fluoxetine, sertraline, paroxetine, citalopram) — Fluoxetine (80mg/day or maximum tolerated dosage) Sertraline (200mg/day or maximum tolerated dosage) Paroxetine (60 mg/day or maximum tolerated dosage) Citalopram (60 mg/day or maximum tolerated dosage)
  Other Names: Prozac; Zoloft; Paxil; Cipramil
  Arms: 2

SUMMARY:
First line treatments fo Obsessive Compulsive Disorder (OCD) are Selective Serotonin Recapture Inhibitors (SSRIs) and Cognitive Behaviour Therapy (CBT) including exposure with response prevention. The aim of the present study is to evaluate the clinical efficacy of GCBT and SSRIs for OCD patients. Other clinical trials have compared these treatments, but with OCD patients without any other psychiatric disorder. In this study patients with current age between 18 and 65 years, with YBOCS score of at least 16 and psychiatric comorbidities will be not excluded. Exclusion criteria will be: OCD secondary to brain trauma, stroke or malformation; current abuse of alcohol or other psychoactive substance, current presence of psychotic symptoms, suicidal risk, psychiatric or clinical comorbidity that might get worse with the medications used in the trial. So, the present study investigates the efficacy of these treatments for a heterogeneous OCD population, trying to identify if the usual treatments are efficient when applied in the public health system that treat not just patients with only OCD diagnosis. Patients will be randomized for GCBT and SSRI, and after treatment will be evaluated by researchers blind to the treatment received.

DETAILED DESCRIPTION:
During the last decades, different pharmacological and psychotherapeutic strategies have been used to treat patients with obsessive compulsive disorder (OCD). Drugs that inhibit the serotonin recapture and the cognitive behavior therapy, that includes the exposure with response prevention and cognitive strategies, have been the most efficient treatment so far. This study's aims are to compare group cognitive-behavior therapy and standard pharmacological treatment (SRIs) in a world real population, using broader inclusion criteria. DSM-IV diagnostic criteria for OCD will be used (APA, 1994) and patients will be interviewed with the following instruments: SCID-I and Y-BOCS. Inclusion criteria are: (1) OCD diagnosis, (2) YBOCS score ≥ 16 (for patients with both obsessions and compulsions) or ≥ 10 (for patients with only obsessions or compulsions), (3) informed consent to participate in this clinical trial. Exclusion criteria are: (1) patients with clinical or neurological diseases that may be worsen by the medications included in treatment protocol, (2) Current substance dependence, (3) Current psychotic symptoms, (4) Current suicide risk. Patients will be randomized in blocks of 12 and with stratification for the following parameters: current SSRI, age, sex and previous response to treatment. Rates of improvement will be based on the results of the YBOCS scores for obsessions and compulsions and on the results of the clinical global impression scale. Pos-treatment measures will be assessed by psychiatrists or psychologists not involved in the patients treatment that will be blind for the treatment being received by the patient. The patient will be considered responsive to treatment when he or she presents a reduction in YBOCS score ≥ 35% of the initial score and a CGI score of 1 (very much improved) or 2 (much improved). The results of this study will help us to identify better health politics planning to a heterogeneous OCD population. So, it will improve our knowledge about the efficacy of the first line treatments in a real world OCD population.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with primary OCD according to the criteria set forth in the DSM-IV;
* Current symptoms causing significant distress (YBOCS score greater than 16);
* Not receiving current adequate treatment;
* Accepting to participate in the study

Exclusion Criteria:

* Having a clinical or neurological disease that might be worsened by the medicines included in the treatment protocol;
* Presenting current substance dependence or abuse;
* Exhibiting current psychotic symptoms; being currently at risk for suicide;
* And, being pregnant or having the intention to become pregnant prior to the end of the treatment protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) (Goodman et al., 1989) and Clinical Global Impressions (CGI) (Guy, 1976) will be implemented at pre and post treatment by a blind evaluator to the treatment received. | 12 weeks

SECONDARY OUTCOMES:
Quality of life measured by SF 36 and social adjustment measured by EAS. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristina B Silva, Psychologist, Principal Investigator — University of Sao Paulo
Locations (1):
- Institute of Psychiatry, Clinics Hospital, University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] da Conceicao Costa DL, Shavitt RG, Castro Cesar RC, Joaquim MA, Borcato S, Valerio C, Miguel EC, Diniz JB. Can early improvement be an indicator of treatment response in obsessive-compulsive disorder? Implications for early-treatment decision-making. J Psychiatr Res. 2013 Nov;47(11):1700-7. doi: 10.1016/j.jpsychires.2013.07.006. Epub 2013 Aug 13. PMID 23948637
- [Derived] Hoexter MQ, Dougherty DD, Shavitt RG, D'Alcante CC, Duran FL, Lopes AC, Diniz JB, Batistuzzo MC, Evans KC, Bressan RA, Busatto GF, Miguel EC. Differential prefrontal gray matter correlates of treatment response to fluoxetine or cognitive-behavioral therapy in obsessive-compulsive disorder. Eur Neuropsychopharmacol. 2013 Jul;23(7):569-80. doi: 10.1016/j.euroneuro.2012.06.014. Epub 2012 Jul 27. PMID 22841131
- [Derived] Belotto-Silva C, Diniz JB, Malavazzi DM, Valerio C, Fossaluza V, Borcato S, Seixas AA, Morelli D, Miguel EC, Shavitt RG. Group cognitive-behavioral therapy versus selective serotonin reuptake inhibitors for obsessive-compulsive disorder: a practical clinical trial. J Anxiety Disord. 2012 Jan;26(1):25-31. doi: 10.1016/j.janxdis.2011.08.008. Epub 2011 Aug 19. PMID 21907540
- [Derived] Fossaluza V, Diniz JB, Pereira Bde B, Miguel EC, Pereira CA. Sequential allocation to balance prognostic factors in a psychiatric clinical trial. Clinics (Sao Paulo). 2009;64(6):511-8. doi: 10.1590/s1807-59322009000600005. PMID 19578654